CLINICAL TRIAL: NCT02022410
Title: Cumulated Ambulation Score and Length of Hospital Stay After TKA
Brief Title: CAS and Length of Hospital Stay After TKA
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Brigitte Jolles, MD, Prof., University of Lausanne Hospitals
Other Study IDs: CHUV 144/13; CAS (Registry Identifier: DAL TKA registry)
Record Dates: First submitted 2013-09-17; First posted 2013-12-27 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: CAS
Keywords: CAS; Length of stay; Rehabilitation localisation; TKA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAS after primary and revision TKA: CAS and RAPT
  Interventions: Other: CAS after primary and revision TKA

INTERVENTIONS:
Other: CAS after primary and revision TKA — CAS and RAPT

SUMMARY:
The purpose of the study is to prospectively evaluate patients who underwent total knee arthroplasty (TKA) using the Cumulated Ambulation Score (CAS)

DETAILED DESCRIPTION:
The number of patients who receive a total knee arthroplasty (TKA) is steadily increasing and although the reliability and the results of this procedure are excellent, intensive functional rehabilitation is needed postoperatively to obtain satisfactory range of motion. Currently, the standard length of stay at our hospital is between 8 and 10 days for patients who undergo TKA.

The length of stay depends not only on factors such as early mobilization, pain management, major or minor complications and logistical or organizational problems (1) (2). It also depends on the availability of adequate services when the patient needs to be transferred to an appropriate facility. Each of these steps can be further developed in order to improve the quality of care for patients, reduce hospital costs and increase the availability of beds (3). As a result, the reduction in average length of stay would not only result in a reduction in cost but also a greater turnover in the number of patients. Several studies show that the application of a post-operative fast-track strategy may reduce the length of stay in a very significant manner with benefit for patients and hospitals (3).Thus, if their condition allows, patients would have rapid post-operative rehabilitation, with early joint mobilization at D0 (operative day) and walking from D1 (the first post-operative day).

The Cumulated Ambulation Score (CAS) (4) is a tool developed and tested for initial predicting the in-patient length of stay following a hip surgery. The CAS consists of documenting the patient's ability and independence while performing 3 basic daily activities (sit to stand, transfer out of bed and mobilization). It is calculated using a score of 0-2 for each parameter, giving a total daily score of 0 to 6 and a score of 0 to 18 during the first 3 post-operative days. The CAS is then the sum of scores of the first 3 post-operative days. This score proves to be an effective tool for predicting the length of stay, and other parameters investigated such as survival rate and return home after a proximal femoral surgery.

ELIGIBILITY:
Inclusion Criteria: Adults after elective TKA -

Exclusion Criteria: No consent form signed, neurological impairment

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TKA patients just after surgery
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
CAS value | The 3rd day after TKA
  Record the CAS values for the first three operative days as mentioned in the protocol

SECONDARY OUTCOMES:
Length of stay | between 4 days and 2 weeks
  Record number of in-hospital days

OTHER OUTCOMES:
Destination at the end of the hospitalisation | at the moment of departure from in-hospital care
  Record the patients' destination at the end of the in-hospital stay: home, rehabilitation centre, residential home or other.

CONTACTS AND LOCATIONS:
Overall Officials: B Jolles, Prof., Study Director — CHUV; Luis C Pereira, MSc, Principal Investigator — CHUV; Georgios Gkagkalis, Dr, Principal Investigator — CHUV
Locations (1):
- CHUV - Hopital Orthopedique, Lausanne, Canton of Vaud, Switzerland